CLINICAL TRIAL: NCT05449054
Title: Continuous Stitches Versus Simple Interrupted Stitches for Anterior Colporrhaphy: Study Protocol for Suture Plication Method: a Randomized Controlled Trial
Brief Title: Continuous Stitches Versus Simple Interrupted Stitches for Anterior Colporrhaphy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christine Bekos, Principan Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sutures in colporrhaphy
Record Dates: First submitted 2022-06-09; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Cystocele; Cystocele, Midline; Vaginal Prolapse; Prolaps Bladder; Pelvic Organ Prolapse
MeSH Terms: conditions — Cystocele; Uterine Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous stitches for anterior colporrhaphy (Active Comparator): Continuous stitches will be used for plication during anterior colporrhaphy. Sutures will be at a distance of no more than 0.5 cm. Trimming of the vagina will be performed if necessary. The anterior vaginal skin is closed with continuous 2/0 vicryl sutures.
  Interventions: Procedure: Anterior colporrhaphy
- Interrupted stitches for anterior colporrhaphy (Active Comparator): Interrupted stitches will be used for plication during anterior colporrhaphy. Sutures will be at a distance of no more than 0.5 cm. Trimming of the vagina will be performed if necessary. The anterior vaginal skin is closed with continuous 2/0 vicryl sutures.
  Interventions: Procedure: Anterior colporrhaphy

INTERVENTIONS:
Procedure: Anterior colporrhaphy — All patients will be operated by the vaginal route. They are prepared under strict aseptic conditions in the dorsal lithotomy position. The bladder is emptied preoperatively with a thin disposable catheter and antibiotic prophylaxis (cefazolin) is administered before incision. A vasoconstricting solution (combination of vasopression and NaCl) is administered and a vertical anterior vaginal incision is made from the apex to two centimeters short of the external urethral meatus using an electric cautery or a scalpel. The vaginal epithelium is grasped on both sides and the fibromuscular layer of the anterior vaginal wall is sharply dissected laterally to the inferior pubic ramus. The bladder is completely dissected from the apex and up to 4 to 6 cm from the pubic ramus. The anterior colporrhaphy is defined as a native tissue repair and rows of absorbable sutures (2/0 vicryl) are used.

SUMMARY:
The anterior vaginal wall is the segment most commonly affected by prolapse. Traditionally, anterior vaginal wall prolapse is repaired via anterior colporrhaphy (native tissue repair), which is known to have a high recurrence rate. Several factors like the suture plication method might affect the outcome of anterior colporrhaphy. The use of single button sutures for example might be associated with the high recurrence rate because the sutures might not be able to retain adequate strength. Nonetheless, no comparative data exist so far regarding the efficacy and safety of anterior colporrhaphy when analyzing the plication method of sutures (= comparison between continuous stiches versus simple interrupted stiches).

The objective of this study is to compare the of patients undergoing anterior colporrhaphy due to symptomatic POP - using either continuous stiches or simple interrupted stiches.

This is a randomized, single-center, superiority trial. Anterior colporrhaphy will be performed in a traditional standardized manner in accordance with the policy of our institution. After midline incision and preparation of vesicovaginal fascia, midline plication of the fibromuscular layer is performed. Patients are randomized either to the group receiving continuous sutures or to the group with simple interrupted stitches. The primary outcome of interest is subjective symptom improvement (evaluated by German version of the pelvic floor questionnaire) assessed at 6 and 12 months after surgery. Secondary outcome variables include anatomical outcomes, condition-specific quality of life and adverse events related to anterior colporrhaphy. Due to the power calculation, an estimated and planned number of participants is 40.

DETAILED DESCRIPTION:
This trial is a single-center, prospective, randomized trial conducted with the aim of determining the superiority of continuous sutures over simple interrupted stitches with regard to the primary outcome in POP patients undergoing anterior colporrhaphy. The study will be a single-blind study, as it is impossible to blind the study surgeon for the surgical procedure to which the subject is assigned. However, all outcome assessors and the subjects will be blinded to the treatment assignment. Postoperative follow-up will take place after 4-6 weeks, 6 months and 12 months. Patients will undergo a standardized urogynecological examination that includes assessment of prolapse with POP-Q measurement. Furthermore subjective outcome will be assessed with standardized questionnaires - our study participants will receive the German version of the pelvic floor questionnaire.

Study setting

This study will be conducted at the urogynecologic outpatient clinic (Division of General Gynecology and Gynecologic Oncology, Department of Obstetrics and Gynecology, Medical University of Vienna). Enrolment, treatment and data collection will be standardized by all sites according to the approved study protocol.

Participants and recruitment

The study population will consist of women aged 18 years or older who are referred to our urogynecologic outpatient clinic due to symptomatic POP. Women with anterior vaginal wall prolapse and an indication for reconstructive pelvic floor surgery - including anterior colporrhaphy with native tissue repair - can be included in this trial.

Intervention

Anterior colporrhaphy will be performed in a traditional and standardized manner in accordance to our surgical policy. Any other concomitant procedures (e.g. vaginal hysterectomy, sacrospinous suspension, superficial perineorrhaphy, posterior recto-vaginal fascia plication, McCall's culdoplasty) will be performed in accordance with each surgeon's preferred technique.

All patients will be operated by the vaginal route. They are prepared under strict aseptic conditions in the dorsal lithotomy position. The bladder is emptied preoperatively with a thin disposable catheter and antibiotic prophylaxis (cefazolin) is administered before incision. A vasoconstricting solution (combination of vasopression and NaCl) is administered and a vertical anterior vaginal incision is made from the apex to two centimeters short of the external urethral meatus using an electric cautery or a scalpel. The vaginal epithelium is grasped on both sides and the fibromuscular layer of the anterior vaginal wall is sharply dissected laterally to the inferior pubic ramus. The bladder is completely dissected from the apex and up to 4 to 6 cm from the pubic ramus. The anterior colporrhaphy is defined as a native tissue repair and rows of absorbable sutures (2/0 vicryl) are used. Depending on preoperative randomization, patients will receive either continuous stitches versus simple interrupted stitches for plication during anterior colporrhaphy. Sutures will be in a distance of no more than 0.5 cm. Trimming of the vagina will be performed if necessary. Anterior vaginal skin is closed with continuous 2/0 vicryl sutures. Participating surgeons will be defined as high volume surgeons in prolapse surgery and will also be part of the urogynecologic core team.

Perioperative management is also standardized and includes preoperative single-shot antibiotics as well as vaginal pack and an indwelling urinary catheter for 24 hours after the surgical procedure.

Patients undergoing anterior with or without apical prolapse correction will have postvoid residual volume measurement at the first postoperative day (when urinary catheter is removed). A postvoid residual volume of 2 x < 100 ml is defined as normal and no further follow- ups are necessary. Postvoid residual volumes of > 150 mL or greater will be considered as abnormal. These patients' volumes will continue mechanical bladder drainage via clean intermittent (self)-catheterisation until the postvoid residual volumes are consistently less than 150 ml. Patients will receive standard analgesic therapy in accordance with the local hospital protocol (Metamizol 1g intravenously, 3 times a day).

Postoperative Management: The patients are instructed to rest for 2 weeks after the operation (not to work, to do sport, to do the cleaning and to carry more than five kilos). They are allowed to return to work after 4 weeks and to take part in sport or have intercourse after 6 weeks. Follow-up visits are scheduled after 4-6 weeks, 6 months and 1 year in our outpatient clinic due to our study protocol. Urogynecological examination is performed at each visit and evaluations are made using the POP-Q measurement system on maximum Valsalva effort in the seated semi-lithotomy position. Objective anatomical cure was defined as a Ba point < -1. Postoperative functional results for symptoms, quality of life and sexuality are evaluated with the Deutsche Beckenboden-Fragebogen. This Pelvic Floor Questionnaire consists of four domains: bladder, bowel, pelvic organ prolapse and sexual function. In every domain various questions assess severity and condition-specific quality of life. Every question is scored on a scale from zero to four. The sum of each individual domain is divided by the maximum reachable score and multiplied by ten, giving a value between zero (0= no symptoms) and ten (10=maximum of symptoms) for each of the domains.

Data collection

At baseline, the following data will be collected: demographics and medical history data (age, body mass index, parity, menopausal and hormone therapy status, current smoking, previous hysterectomy and previous anti-incontinence surgery, and medical comorbidities (diabetes mellitus, connective tissue disorders)), and data from the standardized POPQ examination in a 45° upright sitting position during maximal Valsalva. Patients will be asked to complete the validated questionnaire (Deutscher Beckenboden-Fragebogen).

Scheduled in-person follow-ups will occur at 4 to 6 weeks, 6 and 12 months after the operation. Each check-up will include a clinical examination including POPQ and written questionnaire identical to this at baseline. In addition, an update of current medications, an assessment of new or continuing pelvic floor disorders and adverse events that occurred since the previous evaluation will be obtained by the study coordinator at each visit. All data will be anonymized and collected using case report forms by examiners or trained research coordinators who are blinded to the treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Anterior vaginal wall prolapse beyond the hymen (POPQ point Ba >0) with a central defect.
* Vaginal bulge symptoms
* Reconstructive surgery via native tissue repair is indicated and planned.

Exclusion Criteria:

* Recurrent anterior vaginal wall prolapse
* Anterior vaginal wall prolaps with lateral defect
* Reconstructive surgery using mesh or obliterative surgery is planned
* Known pelvic malignancy
* Current systemic glucocorticoid or immunosuppressant treatment
* Subject is unable or unwilling to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
subjective symptom improvement | 12 months
  differences in the German version of the pelvic floor questionnaire (12 months after the operation compared to preoperative score, ranging from a minimum of 0 (better outcome) to a maximum of 2.875 (worse outcome))

SECONDARY OUTCOMES:
anatomical outcomes | 12 months
  changes in POPQ stages from baseline (stage 0 (no prolapse) to stage 4 (vaginal eversion is essentially complete))
rate of adverse events | 12 months
  differences in intraoperative (bladder injury, ureteral obstruction, massive bleeding) and postoperative (haematoma, vesico-vaginal fistula, ureteral obstruction, urinary tract infection, incomplete bladder emptying, overactive bladder or stress incontinence symptoms, suture erosion, vaginal wound dehiscence, infection or granulation tissue, etc) adverse events
operation time | 1 day
  operation times in minutes
blood loss | 1 day
  intraoperative blood loss in ml
pain killers | 30 days
  postoperative use of pain killers (type of pain killers and dosage)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bodner-Adler, Study Chair — Medical University of Vienna, Department for Obstetrics and Gynecology
Locations (1):
- Medical University of Vienna, Department of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No